CLINICAL TRIAL: NCT02995798
Title: The Characteristics of Regional Bone Quality in the Cervical Vertebrae Considering BMD
Status: Completed | Type: Observational
Sponsor: Gangneung Asan Hospital (Other)
Collaborators: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Moon-Kyu Kim, MD, Ph.D, Professor, Gangneung Asan Hospital
Other Study IDs: Anatomy C-Spine
Record Dates: First submitted 2016-12-09; First posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Cortical Bone Thickness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: T-score ≥-1
  Interventions: Other: Cortical Bone thickness and Hounsfield unit (HU) numbers
- Group B: -2.5<T-score<-1.0
  Interventions: Other: Cortical Bone thickness and Hounsfield unit (HU) numbers
- Group C: T-score≤-2.5
  Interventions: Other: Cortical Bone thickness and Hounsfield unit (HU) numbers

INTERVENTIONS:
Other: Cortical Bone thickness and Hounsfield unit (HU) numbers — Cortical Bone thickness and Hounsfield unit (HU) numbers considering BMD

SUMMARY:
Data of CT images and the femoral neck BMD were obtained from 99 patients who underwent the cervical CT and BMD simultaneously (the gap of both studies was within 6 months) from April 2009 to December 2014. There were 52 females and 47 males. The mean age was 63.7 year (female: 63.4 years, male: 64.1; range 32-86 years). The patient was excluded who had any destructive pathology or severe spondylosis in the cervical pedicle and the cervical lateral mass. Patients were divided into three groups according to femoral neck BMD (Group A, T-score ≥-1; Group B, -2.5<T-score<-1.0; Group C, T-score≤-2.5). Group A had normal BMD patients, Group B had lower normal patients including osteopenic patients and Group C presented osteoporotic patients. The mean HU numbers of cortical bone area in the vertebral canal (cHU, the medial wall of the lateral mass), the posterior wall of transverse foramen (fHU), the medial (mHU), lateral wall (lHU) and trabecular area of pedicle (pHU) were measured on the axial CT images in clinical images.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent the cervical CT and BMD simultaneously (the gap of both studies was within 6 months)

Exclusion Criteria:

* Who had any destructive pathology or severe spondylosis in the cervical pedicle and the cervical lateral mass.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data of CT images and the femoral neck BMD were obtained from 99 patients who underwent the cervical CT and BMD simultaneously (the gap of both studies was within 6 months)
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2009-04; Primary Completion 2014-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Cortical bone Thickness | two weeks
HU number | two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Moon-Kyu Kim, Gangneung, Kangwondo, South Korea

IPD SHARING:
Plan to Share IPD: Undecided